CLINICAL TRIAL: NCT07241962
Title: Prevalence of Hepatitis B and C Within the Chinese Community Residing in Milan
Brief Title: Hepatitis B and C Within the Chinese Community in Milan
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Federica Invernizzi, Doctor, IRCCS Ospedale San Raffaele
Other Study IDs: OBS-CHN-2025
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: HBV (Hepatitis B Virus); HCV Infection
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the effectiveness of targeted screening for Hepatitis B (HBV) and Hepatitis C (HCV) infections in adults aged 18 to 50 from the Chinese community residing in Milan.

The main questions it aims to answer are:

* Does community-based, culturally sensitive screening increase the detection of undiagnosed HBV and HCV infections in this high-risk population?
* What is the level of adherence, satisfaction and awareness regarding rapid testing methods in this community?

Participants will:

* Receive pre-test counseling in Italian or Chinese with the help of an interpreter
* Complete a brief, anonymous questionnaire on demographics, risk factors and awareness of HBV/HCV
* Undergo capillary rapid testing for HBV and/or HCV
* Receive test results during the same visit
* Complete a short post-test satisfaction questionnaire

The study will be conducted in public spaces within Milan's Chinatown, during monthly sessions, until 1,000 participants are enrolled. Each session will last approximately 30-60 minutes per participant.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 50 years
* Self-identified as part of the Chinese community residing in Milan
* Willing and able to provide informed consent
* Willing to undergo HBV and/or HCV rapid screening (capillary blood test)
* Able to complete an anonymous questionnaire on demographics, risk factors and awareness of HBV and HCV infections
* Able to communicate in Italian or Chinese (with interpreter assistance, if needed)

Exclusion Criteria:

* Age under 18 or over 50 years
* Not from the Chinese community or not residing in Milan
* Unable to provide informed consent
* Currently undergoing treatment for HBV or HCV, or with previously confirmed diagnosis of HBV or HCV
* Severe mental or physical illness impairing participation or understanding of consent
* Unable to respond to the questionnaire, even with interpreter assistance
* Pregnant women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 18 to 50 years who self-identify as part of the Chinese community residing in Milan. Participants must be able to provide informed consent, complete a short questionnaire and undergo rapid testing for HBV and/or HCV. Both males and females are eligible. The study aims to reach individuals who may face cultural, linguistic or systemic barriers to healthcare access.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of HBV and/or HCV infections | Day 1 (during the screening session)
  Proportion of participants from the Chinese community residing in Milan who test positive for Hepatitis B surface antigen (HBsAg) and/or anti-HCV antibodies using capillary rapid tests during the screening session

SECONDARY OUTCOMES:
Adherence to rapid HBV/HCV testing | Day 1
  Proportion of participants who complete the full screening process, including pre-test counseling, informed consent, questionnaire and rapid testing
Acceptability of rapid testing methods | Day 1
  Participant satisfaction and perceived acceptability of the capillary rapid testing process, measured through a standardized post-test questionnaire
Demographic profile and risk factors of screened individuals | Day 1
  Distribution of age, sex and self-reported risk factors among participants who undergo screening
Awareness of HBV and HCV infections | Day 1
  Proportion of participants who report prior awareness or knowledge of HBV and/or HCV infections in the pre-test questionnaire